CLINICAL TRIAL: NCT03002272
Title: Transcatheter Aortic Prosthesis Function: A Long-term Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TAVR Durability
Record Dates: First submitted 2016-12-21; First posted 2016-12-23 (Estimated); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TAVR: This observational study will enroll subjects that underwent TAVR more than 3 years ago.
  Interventions: Device: TAVR
- SAVR: Historical controls will be selected from among patients at the same site who underwent isolated bioprosthetic SAVR more than 3 years ago
  Interventions: Device: SAVR

INTERVENTIONS:
Device: TAVR — subjects that underwent TAVR more than 3 years ago
  Groups: TAVR
Device: SAVR — Historical controls will be selected from among patients at the same site who underwent isolated bioprosthetic SAVR more than 3 years ago
  Groups: SAVR

SUMMARY:
In this observational study, the investigators will enroll subjects who underwent TAVR or SAVR more than 3 years ago. Clinical and procedural data from the implant/surgery will be collected, alongside clinical and echocardiographic data from subsequent follow-up visits.

DETAILED DESCRIPTION:
There is limited available information on long term TAVR valve function. In this observational study, the investigators will enroll subjects who underwent TAVR or SAVR more than 3 years ago. Clinical and procedural data from the implant/surgery will be collected, alongside clinical and echocardiographic data from subsequent follow-up visits. Up-to-date echocardiography will be performed and analyzed in a Core Lab to assess valve function yearly.

ELIGIBILITY:
Inclusion criteria for TAVR subjects

a) TAVR performed more than 3 years ago

Exclusion criteria

1. Subjects unable to consent to participate, unless the subject has a legally authorized representative
2. Subjects unwilling to participate
3. Subject has undergone re-intervention to prosthetic aortic valve since TAVR procedure (e.g. balloon valvuloplasty, SAVR, re-do TAVR, paravalvular leak closure)
4. Echocardiographic evidence of prosthetic valve dysfunction within first 3 years post-TAVR (mean aortic gradient ≥20mmHg AND/OR moderate-severe transvalvular aortic regurgitation)

Inclusion criteria for SAVR subjects

1. SAVR performed more than 3 years ago
2. Propensity matched to an enrolled TAVR subject

Exclusion criteria for SAVR subjects e) Subjects unable to consent to participate, unless the subject has a legally authorized representative f) Subjects unwilling to participate g) Subject has undergone re-intervention to prosthetic aortic valve since TAVR procedure (e.g. balloon valvuloplasty, SAVR, re-do TAVR, paravalvular leak closure) h) Echocardiographic evidence of prosthetic valve dysfunction within first 3 years post-SAVR (mean aortic gradient ≥20mmHg AND/OR moderate-severe transvalvular aortic regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational study will enroll subjects that underwent TAVR more than 3 years ago. TAVR.
  Historical controls will be selected from among patients at the same site who underwent isolated bioprosthetic SAVR more than 3 years ago
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Prosthetic valve dysfunction | 7 years
  Mean aortic valve gradient ≥20 mm Hg Moderate-severe transvalvular aortic regurgitation

SECONDARY OUTCOMES:
Change in functional status | discharge from hospital
  Change in functional status from baseline and discharge per NYHA classification
Increase in severity of aortic regurgitation | upto 7 years
  Increase in severity of aortic regurgitation by one or more grading of severity

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No